CLINICAL TRIAL: NCT02352012
Title: A Multi-site Randomized Controlled Study of Interventional Treatment of Refractory Pneumothorax by Bronchoscope
Brief Title: Interventional Treatment of Refractory Pneumothorax by Bronchoscope
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Collaborators: Changhai Hospital (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Second Affiliated Hospital of Third Military Medical University (Other); China Meitan General Hospital (Other); Micro-Tech (Nanjing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: tdhx007; 201402024007 (Other Grant/Funding Number: 201402024)
Record Dates: First submitted 2014-11-18; First posted 2015-01-30 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Pneumothorax
Keywords: Interventional Treatment; Refractory Pneumothorax; Bronchoscope
MeSH Terms: conditions — Pneumothorax | interventions — Blood Transfusion, Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Autologous blood group A (Experimental): Autologous blood was perfused to the target pulmonary segment
  Interventions: Other: Autologous blood
- Bronchial plug group B (Experimental): Bronchial plug was placed to the target pulmonary segment
  Interventions: Device: Bronchial plug
- control group (No Intervention): Control group was given to continuous negative pressure drainage

INTERVENTIONS:
Other: Autologous blood — Autologous blood was perfused to the target pulmonary segment
  Arms: Autologous blood group A
Device: Bronchial plug — Bronchial plug was placed to the target pulmonary segment
  Arms: Bronchial plug group B

SUMMARY:
The purpose of this study is to determine whether injecting autologous blood or putting bronchial plug through bronchoscope is effective in the treatment of refractory pneumothorax.

DETAILED DESCRIPTION:
This is a multi-site, controlled, randomized study. Refractory pneumothorax is a challenge for respiratory physicians. Many patients present recurrent pneumothorax. Thoracic closed drainage is a basic and effective treatment to pneumothorax. Chronic obstructive pulmonary disease(COPD)is one of the main causes of spontaneous pneumothorax. Many patients precluded the performance of surgery for poor pulmonary function. In China, economical load is another reason for patients who are unwilling to surgery. So we want to seek a cheap, effective and safe method for refractory pneumothorax. We will adopt three methods in this study. Conventional thoracic closed drainage was continuously used in the control group, autologous blood was perfused to the target pulmonary segment in the treatment A group and self-made silicone bronchial plug was placed to the target pulmonary segment in the treatment B group. The leak position was detected by biliary lithotomy balloon. Main outcome measures: duration of continuous leakage. Secondary end-points included the lung reexpanded, hospital costs and hospital stays etc.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous pneumothorax has been treating with thoracic closed drainage for 7 days, the patient has still persistent air leakage;
* Patients informed consent to participate in this study and can complete the requirements of the follow-up visit

Exclusion Criteria:

* Patients with severe abnormal gas exchange are defined as PaCO2>50mmHg(6.6kPa) or PaO2<45mmHg(6.0kPa) ;
* Patients have systemic disease or cancer which affect the survival time ;
* Patients have other serious diseases (the researchers think patient is not an appropriate candidate) which affect the evaluation or follow-up in research;
* Patients are not suitable for or unable to tolerate bronchoscopy procedures;
* Patients have active tuberculosis;
* Patients have any disease or condition that interferes with completion of initial or follow-up assessments of the effectiveness endpoints including interference test of nerves or skeletal muscle disease;
* Patients have demonstrated unwillingness or inability to complete screening or baseline data collection procedures;
* Patient participated in a study of an investigational drug or device within the past 30 days prior to participation in this study, or is currently participating in another clinical study;
* Female patient of childbearing potential has a positive result from a pregnancy test.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-02 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Duration of air leakage | up to two weeks

SECONDARY OUTCOMES:
duration of pulmonary atelectasis | up to two weeks

OTHER OUTCOMES:
Arterial blood gas | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
complications | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Complications refers to the complications related to bronchoscopy treatment(include hemoptysis, short of breath, chest pain, fever )
hospital costs | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
Duration of hospital stays | participants will be followed for the duration of hospital stay, an expected average of 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Faguang Jin, MD & PhD, Principal Investigator — Tang-Du Hospital
Locations (1):
- Tangdu Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Gilbert CR, Toth JW, Osman U, Reed MF. Endobronchial valve placement as destination therapy for recurrent pneumothorax in the setting of advanced malignancy. Respir Care. 2015 Mar;60(3):e46-8. doi: 10.4187/respcare.03540. Epub 2014 Oct 21. PMID 25336533
- [Background] Cundiff WB, McCormack FX, Wikenheiser-Brokamp K, Starnes S, Kotloff R, Benzaquen S. Successful management of a chronic, refractory bronchopleural fistula with endobronchial valves followed by talc pleurodesis. Am J Respir Crit Care Med. 2014 Feb 15;189(4):490-1. doi: 10.1164/rccm.201311-1965LE. No abstract available. PMID 24528320
- [Background] Yamashita T, Urabe N. [Prolonged iatrogenic pneumothorax with refractory hepatic hydrothorax treated successfully with local anesthetic thoracoscopic talc poudrage]. Kyobu Geka. 2013 Jun;66(6):460-3. Japanese. PMID 23917049
- [Background] Odaka M, Akiba T, Mori S, Asano H, Yamashita M, Kamiya N, Morikawa T. Thoracoscopic surgery for refractory cases of secondary spontaneous pneumothorax. Asian J Endosc Surg. 2013 May;6(2):104-9. doi: 10.1111/j.1758-5910.2012.00161.x. Epub 2012 Oct 29. PMID 23107020
- [Background] Iyama S, Sato T, Murase K, Kikuchi S, Kamihara Y, Ono K, Takada K, Miyanishi K, Sato Y, Takimoto R, Kobune M, Obama T, Miyajima M, Watanabe A, Higami T, Hirayama Y, Kato J. Successful treatment by fibrin glue sealant for pneumothorax with chronic GVHD resistant to autologous blood patch pleurodesis. Intern Med. 2012;51(15):2011-4. doi: 10.2169/internalmedicine.51.7355. Epub 2012 Aug 1. PMID 22864128
- [Background] Lin XM, Liu Y, Chi C, Lin CX, Yang Y. Efficacy of an absorbable polyglycolic acid patch in surgery for pneumothorax due to silicosis. J Cardiothorac Surg. 2012 Mar 6;7:18. doi: 10.1186/1749-8090-7-18. PMID 22394587
- [Background] Lin XM, Lin CX, Chi C. [Application of absorbable Neoveil patch in operation on refractory pneumothorax in silicosis patients]. Zhonghua Lao Dong Wei Sheng Zhi Ye Bing Za Zhi. 2010 Jan;28(1):60-1. No abstract available. Chinese. PMID 20426989
- [Background] Bialas RC, Weiner TM, Phillips JD. Video-assisted thoracic surgery for primary spontaneous pneumothorax in children: is there an optimal technique? J Pediatr Surg. 2008 Dec;43(12):2151-5. doi: 10.1016/j.jpedsurg.2008.08.041. PMID 19040924
- See also: Click here for more information about this study: different treatment methods for different causes of pneumothorax — http://www.ncbi.nlm.nih.gov/pubmed